CLINICAL TRIAL: NCT06890156
Title: Bridging Gaps and Scaling Up: a School Readiness Programme for Child-parent-teacher Triad in Bangladesh, Nepal and Tanzania
Brief Title: Every Newborn Reach Up Early Education Intervention for All Children Education (ENREACH) Education
Acronym: ENREACH-ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); University of Glasgow (Other); London School of Hygiene and Tropical Medicine (Other); Golden Community, Nepal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR-24085; 110505-001. (Other Grant/Funding Number: International Development Research Centre (icddr,b))
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: School Readiness; School Environment
Keywords: School readiness; Early childhood care and education (ECCE); Early childhood development (ECD); Pre-primary education; disabilities; Cluster randomized controlled trial (cRCT)

STUDY DESIGN:
Intervention Model Description: Prior to enrolling study participants, we will conduct sensitization meetings with each selected government primary school. These meetings will be oriented toward community leaders, caregivers of children with or without disabilities, and SMCs to introduce them to the programme, ensure the inclusion of all children, and address concerns related to gender, poverty, and disability.
  A disability-inclusive module will be delivered to preschoolers in their regular pre-primary classrooms by trained pre-primary teachers. This module will cover foundational skills, the importance of play, communication, socio-emotional learning, and strategies for adapting the curriculum to accommodate children with disabilities.
  Additionally, the ENREACH parent group school readiness intervention package will be provided to parents during monthly parent-teacher meetings, facilitated by trained preschool teachers.
Who Masked: Outcomes Assessor
Masking Description: All assessors will be blinded to the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Intervention (Active Comparator): Caregivers and their pre-school children aged 48-84 months, enrolled in pre-primary education.
  Interventions: Behavioral: ENREACH child-parent-teacher triad
- Arm 2: Control (No Intervention): Caregivers and their children aged 48-84 months, enrolled in pre-primary education.

INTERVENTIONS:
Behavioral: ENREACH child-parent-teacher triad — Prior to enrolling study participants, we will conduct sensitization meetings with each selected government primary school. These meetings will be oriented toward community leaders, caregivers of children with or without disabilities, and school management committees to introduce them to the program, ensure the inclusion of all children, and address concerns related to gender, poverty, and disability.
  A disability-inclusive module will be delivered to preschoolers in their regular pre-primary classrooms by trained pre-primary teachers. This module will cover foundational skills, the importance of play, communication, socio-emotional learning, and strategies for adapting the curriculum to accommodate children with disabilities.
  ENREACH parent group school readiness intervention package will be provided to parents during monthly parent-teacher meetings, facilitated by trained preschool teachers.
  Arms: Arm 1: Intervention

SUMMARY:
The goal of the project is to assess the scale-up of the program, focusing on improving school readiness among preschool children, enhancing capacity building for parents and teachers, and utilizing a cluster randomized controlled trial (cRCT). The primary research questions are to seek answer-

* What specific adaptations are necessary for an innovative, disability-inclusive early education training program to become a fully inclusive model that enhances teachers' engagement and practices in pre-primary classrooms in Nepal, Tanzania, and Bangladesh?
* How can a new, equitable 'School Readiness Programme for the child-parent-teacher triad' be effectively scaled within national government pre-primary platforms using a cRCT?
* How can the outcomes of the 'School Readiness Programme for the child-parent-teacher triad' be implemented in a cost-effective manner by key stakeholders across the three sites?

The research will examine an adapted inclusive early education training programme will lead to improved teaching practices, enhanced parental capacity, and better school readiness for all children compared to standard education programme; and b) the child-parent-teacher triad model can be scaled effectively within the government primary education systems.

DETAILED DESCRIPTION:
In Bangladesh, Multiple Indicator Cluster Survey shows that only 18.9% of children aged 3-5 attend early childhood care and education (ECCE) programmes, and 25.5% are not developing at the expected rate (Bangladesh Bureau of Statistics and UNICEF, 2019). In Nepal, there are 35,991 early childhood development (ECD) and ECCE centers, unevenly distributed due to geographical barriers, with a very low enrollment (0.21%) of children with disabilities. Similarly, in Tanzania, efforts to ensure inclusive education in pre-primary schools face challenges with attendance and funding for disability schools in ECCE (Davis, D., et al, 2021).

Despite ongoing efforts through ECCE programmes to promote effective school readiness globally, there exists a considerable and enduring gap in both the access to and quality of ECCE programmes for all children across three countries. This knowledge gap is rooted in the intersectionality of barriers affecting school readiness and scaling up.

This project builds on previous successful work in Bangladesh, Nepal and Tanzania, that focused on the readiness of both children and caregivers to enter the preschool education programme, through an initiative called Every Newborn-Reach Up Early Education Intervention for All Children (ENREACH) (Miah et al, 2024). This new applied research will support the adaptation of the ENREACH programme to incorporate key components on teacher readiness to facilitate a seamless transition to pre-primary education. The justification behind this innovation lies in incorporating key components of teacher readiness into the ENREACH programme, positioning it as an ideal and promising solution for bridging gaps to greater inclusion and increasing opportunities to scaling up across three countries

Objectives:

Objective 1:

To enhance teacher engagement and teaching practices by adapting an innovative disability-inclusive early education training programme into a fully inclusive programme that involves children, parents, teachers and the community.

Objective 2:

Generating knowledge on factors that can facilitate the scaling of the child-parent-teacher triad innovation, including cost-effectiveness.

Objective 3:

To mobilize the key stakeholders within the educational systems under the Ministry of Education in all 3 countries, on the basis of programme results to improve policy and practice to transfer into a government supported programmes.

Study design This study will employ a cluster (sub-districts/wards/municipalities) randomized controlled trial (cRCT) with an embedded qualitative component. It will evaluate scale-up strategies, emphasizing teachers' capacity for preschool to early primary education transition and parents' ability to improve children's school readiness.

Study settings The ENREACH ED study will be conducted at Kushtia and Gaibandha districts in Bangladesh and at Dhading and Nuwakot in Nepal and at Temeke and Kigamboni in Tanzania.

Methods by Objectives Objective 1: ADAPTATION

Step 1: The investigators will refine the tested ENREACH parenting pre-school readiness package by incorporating the following areas:

A) Revise the Pre-school Readiness Parenting Package to ensure it is also aligned to pre-school teacher-pedagogy: the investigators aim to enhance the ENREACH pre-school parenting package by incorporating pre-academic foundational skills and play-based activities, fostering holistic skills development. This includes creating an inclusive environment, promoting play-based learning, storytelling, pre-reading, pre-numeracy skills, drawing, writing, and supporting socio-emotional needs. Collaboration with Ministry of Education representatives and development partner, like the World Bank, ensures alignment with each country's ECCE policy and early learning standards.

B) Develop a teacher training manual: A training module for pre-primary education (PPE)/ECD teacher training, will be developed to promote pre-school teachers' skills in ECCE. These will include foundational skills, importance of play, communication, socio-emotional learning and ways to adapt the curricula for children with disabilities. The content, standards, framework, and pathways will be customized in collaboration with expert educational stakeholders in these settings.

C) Develop a Community Stakeholder Awareness Package: An additional Information Education and Communication (IEC) package including leaflet, poster and short videos will be developed specifically to sensitize key stakeholders including, PPE/ECD teachers, caregivers of children with disabilities, the community leaders and School Management Committee (SMC) about ENREACH ED programme.

Target participants:

Teachers: The teacher training initiative will involve a total of 24 PPE/ECD teachers and 24 headmasters evenly distributed among 24 intervention schools in each country. Upon the completion of the intervention programme, the investigators will extend training to 144 teachers and headmasters in the control group to facilitate the implementation of the programme with government support across three countries.

Parent-child dyad: The study will encompass 3000 caregivers of children from 144 government primary school (GPS)/ECD centres (72 GPS/ECD centres for intervention and 72 control) across two districts in each country.

Outcome variables: Anticipated primary outcome is improved children's school readiness. Secondary outcomes are enhanced parental knowledge, attitudes and practice for school readiness, parent's mental health, children's quality of life, increased teachers' competence, home environment and better school environment.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 48-84 months
* Enrolled in preschools
* Residing in the catchment areas of GPS
* Include/over sample for children with functional disabilities even if they are over 84 months of age.

Exclusion Criteria:

* Un-consenting parents
* Intervention school of EN-REACH study

Ages: 48 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Measuring Early Learning Quality and Outcomes (MELQO) | 40 Minutes
  School readiness (per-literacy, numeracy, executive functions, and social-emotional learning) will be assessed using the Measuring Early Learning Quality and Outcomes (MELQO)

SECONDARY OUTCOMES:
Early childhood version of Home Observation for Measurement of Environment | 30 Minutes
  To measure the quality of home stimulation
Pediatric Quality of Life Inventory (PedsQL) | 30 Minutes
  Physical functioning, emotional functioning, social functioning
Measure of Early Learning Environment (MELE) | 90 minutes
  School Environment
Feeling Questionnaires | 5 minutes
  Depression
Teacher Interview Report | 20 minutes
  Competency
Knowledge and Practice questionnaire | 30 minutes
  To assess knowledge and practices regarding school readiness
Anthropometry | 5 minutes
  Height, Weight
Washington/UNICEF child functioning | 20 minutes
  It assess multiple functional difficulties, such as vision, hearing, mobility, self-care, communication, learning, memory, emotional wellbeing (anxiety, depression), behavior problem, attention, routine changes, and social interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Jena Derakhshani Hamadani, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
The investigators have a six-year track record of equitable partnership between sites (Nepal, Bangladesh, Tanzania and London School of Hygiene & Tropical Medicine) with data sharing agreements already in place. The data will be owned by each country institution and pooled data by the study team. We have already established small committees which include the Principle Investigator (PI) and each site PI who will review any requests for data beyond the original team e.g. - Doctorate of Philosophy formal data sharing agreements will be signed by both parties. However, we will not share any identifiable related individual participant data with other researchers.
Supporting Information: SAP
Time Frame: From December 2025 until analysis is completed A
Access Criteria: All the PIs of each site and statisticians

REFERENCES:
- [Background] Davis, D., Miller, D., Mrema, D., Matsoai, M., Mapetla, N., Raikes, A., & Burton, A. (2021). Understanding perceptions of quality among early childhood education stakeholders in Tanzania and Lesotho: A multiple qualitative case study. Social Sciences & Humanities Open, 4(1), 100153.
- [Background] Miah MAA, Chandna J, Gurung R, Masoud NS, Paul P, Ameen S, Basnet O, Miraji M, Tann C, Mili IA, Hossain AKMT, Chowdhury AI, Alam A, Milner KM, Arifeen SE, Kc A, Manji K, Lynch P, Lawn JE, Hamadani JD; EN-REACH collaborative group. Every Newborn-Reach Up Early Education Intervention for All Children (EN-REACH)- a parent group intervention for school readiness in Bangladesh, Nepal, and Tanzania: study protocol for a cluster randomized controlled trial. Trials. 2024 Aug 23;25(1):556. doi: 10.1186/s13063-024-08381-6. PMID 39180108
- [Background] Bangladesh Bureau of Statistics (BBS) and UNICEF, Multiple Indicator Cluster Survey-2019. 2019